CLINICAL TRIAL: NCT02739633
Title: Phase II Study of Weekly Genexol®-PM Plus Gemcitabine in Subjects With Recurrent and Metastatic Adenocarcinoma of the Pancreas
Brief Title: Study of Weekly Genexol®-PM Plus Gemcitabine in Subjects With Recurrent and Metastatic Adenocarcinoma of the Pancreas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Genexol-PM PC
Record Dates: First submitted 2016-03-21; First posted 2016-04-15 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Recurrent Adenocarcinoma of the Pancreas; Metastatic Adenocarcinoma of the Pancreas
Keywords: Chemotherapy; Gemcitabine; Recurrent and metastatic adenocarcinoma of the pancreas; Genexol-PM; Paclitaxel
MeSH Terms: conditions — Recurrence | interventions — genexol-PM; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Genexol-PM + Gemcitabine (Experimental): Genexol-PM125 mg/m2 will be administered in combination with gemcitabine 1,000 mg/m2 weekly for 3 weeks followed by one week of rest. Each cycle is 28 days.
  Interventions: Drug: Genexol-PM; Drug: Gemcitabine

INTERVENTIONS:
Drug: Genexol-PM — 125 mg/m2 given intravenously over 60 minutes for 3 weeks (days 1, 8 and 15) with 1 week rest. Patients will continue until they experience disease progression or significant toxicity.
  Other Names: Cremorphor EL-free paclitaxel
Drug: Gemcitabine — 1000 mg/m2 given intravenously for 3 weeks (days 1, 8 and 15) with 1 week rest. Patients will continue until they experience disease progression or significant toxicity.

SUMMARY:
Phase II Study of Weekly Genexol®-PM Plus Gemcitabine in Subjects With Recurrent and Metastatic Adenocarcinoma of the Pancreas.

DETAILED DESCRIPTION:
The aim of the this phase II study is to assess the efficacy and safety of a combination treatment of Genexol®-PM plus gemcitabine in patients with recurrent and metastatic adenocarcinoma of the pancreas.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has definitive histologically or cytologically confirmed recurrent and metastatic adenocarcinoma of the pancreas. The definitive diagnosis of recurrent and metastatic pancreatic adenocarcinoma will be made by integrating the histopathological data within the context of the clinical and radiographic data. Patients with islet cell neoplasms are excluded.
2. Initial diagnosis of recurrent and metastatic disease must have occurred ≤6 weeks prior to randomization in the study.
3. Patient has one or more lesions measurable by CT scan or MRI (if patient is allergic to CT contrast media).
4. Male or non-pregnant and non-lactating female, and ≥ 20 years of age.
5. Patient must meet the following blood counts at Baseline (obtained ≤14 days prior to randomization):

   * Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L
   * Platelet count ≥ 100,000/mm3 (100 × 10^9/L)
   * Hemoglobin (Hgb) ≥ 9 g/dL.
6. Patient has the following blood chemistry levels at Baseline (obtained ≤14 days prior to randomization):

   * AST (SGOT), ALT (SGPT) ≤ 2.5 × upper limit of normal range (ULN), unless liver metastases are clearly present, then ≤ 5 × ULN is allowed.
   * Total bilirubin ≤ULN
7. Patient has a Karnofsky performance status (KPS) ≥ 70. Two observers will be required to assess KPS. If discrepant, the one with the lowest assessment will be considered true.
8. Patient has voluntarily agreed to participate in the study, and signed the Informed Consent Form (ICF) prior to participation in any study-related activities.

Exclusion Criteria:

1. History of malignancy in the last 5 years. Patients with prior history of in situ cancer or basal or squamous cell skin cancer are eligible. Patients with other malignancies are eligible if they were cured by surgery alone or surgery plus radiotherapy and have been continuously disease-free for at least 5 years.
2. Patients have uncontrolled bacterial, viral, or fungal infections
3. Patient has known historical or active infection with HIV, hepatitis B, or hepatitis C.
4. Patients have a history of allergy or hypersensitivity to any of Paclitaxel, Gemcitabine, or Cremophor EL.
5. Patients with high cardiovascular risk, including recent coronary stenting or myocardial infarction in the past 6 months.
6. History of Peripheral Artery Disease (e.g,. claudication, Leo Buerger's disease).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) as assessed by RECIST. | 8 weeks
  ORR will be summarized as the percentage of participants who achieved a confirmed complete (CR) or partial response (PR) using RECIST guidelines.
  Response is confirmed at least 4 weeks later.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 2 years
  Time from the date of enrollment until the date of objective disease progression or the date of death.
  PFS will be summarized using Kaplan-Meier methods.
Overall survival (OS) | 2 years
  OS will be summarized using Kaplan-Meier methods.
Disease control rate (DCR) | 8 weeks
  DCR is defined as the percentage of patients who have achieved complete response, partial response and stable disease
Number of participants with adverse events | Baseline up to Day 21 after the last dose of study treatment
  A adverse event (AE) is as any AE occurring or worsening on or after the first treatment of any study drug, and within 21 days after the last dose of the last study drug.
  Severity grades according to NCI CTCAE version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Woo Lee, M.D., Principal Investigator — Ajou University Medical Center
Locations (1):
- Samyang Biopharmaceuticals, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No